CLINICAL TRIAL: NCT00426829
Title: Phase I Study of Proton Radiotherapy and Bevacizumab for Primary Liver Tumors
Brief Title: Proton Therapy and Bevacizumab for Primary Liver Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low Accural
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0881
Record Dates: First submitted 2007-01-23; First posted 2007-01-25 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma; Cholangiocarcinoma
Keywords: Liver Cancer; Biliary Tract; Hepatocellular Carcinoma; Cholangiocarcinoma; Bevacizumab; Proton Therapy; Radiation Therapy; PT; RT; Proton RT; Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Bevacizumab; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proton Therapy + Bevacizumab (Experimental): Proton Therapy + Bevacizumab
  Interventions: Drug: Bevacizumab; Radiation: Proton Radiation Therapy

INTERVENTIONS:
Drug: Bevacizumab — 10 mg/kg by vein every 14 days +/- 2 days, starting on day 1.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Radiation: Proton Radiation Therapy — 3 Gy dose/fraction x 20 fractions.
  Other Names: PT; RT; Proton RT

SUMMARY:
Primary Objectives:

1. To evaluate the safety of the treatment of patients with technically or medically inoperable hepatocellular carcinoma and cholangiocarcinoma with proton therapy and concurrent bevacizumab biotherapy.
2. To identify the maximum tolerated dose (MTD) using this combination.

Secondary Objectives:

1. To evaluate local control rate within the radiation field, hepatic control rate outside the treatment field, time to radiographic progression and 2 year survival rate.
2. To analyze dose-volume characteristics that influence the development of radiation induced liver disease (RILD) and GI bleeds that may occur.
3. To assess quality of life during and after chemoradiation therapy.

DETAILED DESCRIPTION:
Proton beams are designed to deliver a high dose of radiation to the abnormal tissues while sparing surrounding normal tissues. Bevacizumab is a biotherapy that is designed to prevent or slow down the growth of cancer cells by blocking the growth of blood vessels.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete physical exam. Blood (about 2 tablespoons) and urine will be collected for routine tests. You will have chest x-rays and a computed tomography (CT) scan of your abdomen (stomach area) and pelvis. Women who are able to have a children must have a negative urine pregnancy test.

You will then have a radiation treatment planning session called a simulation. You will get a CT scan of your abdomen, and marks will be placed on your skin to help guide the radiation treatments when you return for the actual treatments. At around the same time, you will receive your first dose of bevacizumab through a needle in your vein. The infusion will at first last 90 minutes. If there are no allergic reactions, fevers, or chills, the infusion will be shortened to 60 minutes and then 30 minutes for later infusions. Your second dose of bevacizumab will be given with the start of radiation therapy treatments. Your final dose of bevacizumab will be given 2 weeks later. You will receive radiation therapy once a day, for 5 days in a row (Monday-Friday) for 4 weeks (total of 20 treatments).

During this study, you will have physical exams weekly during treatment, 1 month after the last proton beam therapy visit and then every 3 months thereafter. Every week, while receiving proton beam therapy, blood (about 2 teaspoons) will be drawn to check for any side effects. You will be asked about any side effects you may be experiencing.

You may remain on study for as long as you are benefitting. You will be taken off study if the disease gets worse or intolerable side effects occur.

After participation in this study is over, you will have follow-up evaluation every 3 months for 2 years. During these visits, you will have a physical exam. You will have CT scans. Blood (about 2 teaspoons) will be drawn for routine tests.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of metastatic colon cancer. The use of bevacizumab with proton beam therapy is investigational. Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of primary liver cancer (hepatocellular carcinoma or cholangiocarcinoma). Patients with non-metastatic, unresectable disease are eligible. Patients with positive margins after surgical resection are eligible. Metastasis is defined as unequivocal evidence of extrahepatic disease based on CT imaging, excluding nodal disease.
* Tumors must not be greater than 10cm (small satellite lesions around a larger lesion are allowed), all of which can be encompassed in a radiation treatment field (as assessed by the radiation oncologist).
* Prior chemotherapy, transarterial chemoembolization and radiofrequency ablation are permitted. A minimum of four weeks must have elapsed between prior treatment and planned protocol therapy.
* Prior liver resection is permitted as long as the interval between surgery and enrollment is at least 4 weeks.
* Karnofsky performance status >/= 70 are eligible.
* There is no age restriction.
* Absolute granulocyte count >/= 1,500 cells/mm3, hemoglobin >/= 8 gm/dL and platelet count >/= 80,000 cells/mm3.
* Serum creatinine </= 1.5 mg/dl.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) </= 3 times the upper limit of normal. Serum bilirubin </= 5mg/dL prior to the start of therapy.
* A signed study-specific consent form, which is attached to this protocol.

Exclusion Criteria:

* Child-Pugh class C cirrhosis.
* Gross ascites seen on CT that precludes accurate targeting of the tumor with radiation therapy
* Proteinuria at screening as demonstrated by either Urine protein:creatinine (UPC) ratio > 1.0 at screening OR Urine dipstick for proteinuria > 2+ (patients discovered to have > 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate < 1g of protein in 24 hours to be eligible).
* Patients currently receiving anticoagulation treatment with coumadin, low molecular weight heparin or IV heparin. Evidence of bleeding diathesis or coagulopathy. Anticoagulation for line maintenance is permitted.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study; fine needle aspirations or core biopsies within 7 days prior to Day 0.
* Serious, nonhealing wound, ulcer, or bone fracture.
* Clinically significant cardiac disease (e.g., uncontrolled hypertension [blood pressure of >150/100 mmHg on medication], history of myocardial infarction within 6 months, unstable angina), New York Heart Association (NYHA) Class II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or Class II or greater peripheral vascular disease.
* History of aneurysms, strokes, transient ischemic attacks, and arteriovenous malformations within 6 months.
* Prior unanticipated severe reaction to bevacizumab.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Patients who have had an organ allograft.
* Pregnant women are excluded from this study; women of childbearing potential must agree to practice adequate contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) and to refrain from breast feeding, as specified in the informed consent. Women of child-bearing potential are defined as those women who have not had surgical sterilization or been menopausal for 12 consecutive months.
* Male patients must agree not to father a child and must agree to use a condom.
* Prior radiation therapy to an upper abdominal or lower thoracic field that could overlap with the proposed treatment field.
* Serious concomitant medical or psychiatric disorders that place the patient at high risk for non-compliance with or morbidity due to protocol therapy.
* Patients with a history of hypertension must be well-controlled (</= 140/90 mmHg on a stable regimen of antihypertensive therapy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Toxicity (during and within 1 month after completion of radiotherapy) | 1 month +/- 1 week upon completion of concurrent chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Krishnan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T. M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zhang X, Li G, Li X, Liang Z, Lan X, Mou T, Xu Z, Fu J, Wu M, Li G, Wang Y. Effect of single-incision plus one port laparoscopic surgery assisted with enhanced recovery after surgery on colorectal cancer: study protocol for a single-arm trial. Transl Cancer Res. 2021 Dec;10(12):5443-5453. doi: 10.21037/tcr-21-1361. PMID 35116390
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org